CLINICAL TRIAL: NCT02405637
Title: Enteral Administration of a Simulated Amniotic Fluid In Preventing Feeding Intolerance And Necrotizing Enterocolitis In Very Low Birth Weight Neonates
Brief Title: Simulated Amniotic Fluid In Preventing Feeding Intolerance and Necrotizing Enterocolitis VLBW Neonates
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rania Ali El-Farrash (Other)
Responsible Party: Sponsor-Investigator, Rania Ali El-Farrash, Enteral Administration of a Simulated Amniotic Fluid In Preventing Feeding Intolerance And Necrotizing Enterocolitis In Very Low Birth Weight Neonates, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU 7/2013
Record Dates: First submitted 2015-02-23; First posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Necrotizing Enterocolitis
Keywords: Feeding intolerance; Simulated amniotic fluid; Necrotizing enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SAFE group (Experimental): simulated amniotic fluid 20cc/kg/day enterally divided according to number of feds (syringe for every fed). This amount provides enteral 4.5μg rhG-CSF / kg/day and enteral 88IU rhEPO / kg/day.
  Interventions: Drug: simulated amniotic fluid 20cc/kg/day enterally
- placebo (Placebo Comparator): distilled water 2.5 ml/kg every 3 hours enterally
  Interventions: Drug: distilled water

INTERVENTIONS:
Drug: simulated amniotic fluid 20cc/kg/day enterally — simulated amniotic fluid 20cc/kg/day enterally for a maximum of 7 days.
  Other Names: SAFE solution
  Arms: SAFE group
Drug: distilled water — distilled water 20 ml/kg/day for maximum of 7 days.
  Arms: placebo

SUMMARY:
The human fetus swallows over 200 ml of amniotic fluid per kilogram of weight each day and such swallowing is essential for normal small bowel development.Growth factors found in the amniotic fluid have been shown to promote proliferation of fetal intestinal cells. As feeding intolerance is a common problem among premature neonates, the investigators will study the role of enteral administration of simulated amniotic fluid solution in prevention of feeding intolerance and NEC in premature neonates.

DETAILED DESCRIPTION:
Very Low Birth Weight (VLBW) neonates.

Participants will be followed for the duration of hospital stay until discharge or death.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants with birth weight 1.5 Kg

Exclusion Criteria:

* Congenital or acquired anomaly of the gastrointestinal tract (i.e., omphalocele, tracheoesophageal fistula, intestinal perforation).
* Other major congenital anomalies (congenital heart disease, neural tube defect, congenital diaphragmatic hernia, trisomy, etc.).

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Necrotizing enterocolitis by modified Bell criteria, mortality in percentage, hospital stay in days. The outcome measure will be assessed within 2 months | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rania A El-Farrash, MD, Study Director — ASU
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt